CLINICAL TRIAL: NCT05330689
Title: How Does Platelet Dose Impact Clinical Outcomes After PRP Treatment?
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding for study equipment
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Leon Scott, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRPTreatment
Record Dates: First submitted 2022-04-09; First posted 2022-04-15 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Osteoarthritis, Knee; Arthritis; Platelet rich plasma
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Arthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Sample group 1 (Active Comparator): Sample of subjects with primary osteoarthritis of the knee
  Interventions: Biological: PRP injection dose (<5 billion platelets)
- Sample group 2 (Active Comparator): Sample of subjects with primary osteoarthritis of the knee
  Interventions: Biological: PRP injection dose (between 5 and <10 billion platelets)
- Sample group 3 (Active Comparator): Sample of subjects with primary osteoarthritis of the knee
  Interventions: Biological: PRP injection dose (between 10 and <20 billion platelets)
- Sample group 4 (Active Comparator): Sample of subjects with primary osteoarthritis of the knee
  Interventions: Biological: PRP injection dose (20 billion or greater platelets)
- Sample group 5 (Placebo Comparator): Sample of subjects with primary osteoarthritis of the knee
  Interventions: Other: Saline injection control

INTERVENTIONS:
Biological: PRP injection dose (<5 billion platelets) — PRP injection with a dose of platelets that is less than 5 billion platelets
  Arms: Sample group 1
Biological: PRP injection dose (between 5 and <10 billion platelets) — PRP injection with a dose of platelets that is between 5 and <10 billion platelets
  Arms: Sample group 2
Biological: PRP injection dose (between 10 and <20 billion platelets) — PRP injection with a dose of platelets that is between 10 and <20 billion platelets
  Arms: Sample group 3
Biological: PRP injection dose (20 billion or greater platelets) — PRP injection with a dose of platelets that is 20 billion platelets or greater
  Arms: Sample group 4
Other: Saline injection control — Saline control
  Arms: Sample group 5

SUMMARY:
The purpose of this study is to determine which platelet rich plasma (PRP) injection dosage provides the most improvement in a patient's knee pain level at 26 weeks post-injection.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a chronic progressive disease affecting more than 20% of people older than 45 years. A myriad of different treatments have been proposed in the scientific literature, and current treatment options include conservative and surgical procedures in which the main objective is to relieve pain and improve function.

Conservative nonsurgical interventions include weight management, physical therapy, analgesics, nonsteroidal anti-inflammatory drugs (NSAIDS), corticosteroid and hyaluronic acid injections. Although these agents have been beneficial in the short term, there is a lack of evidence that such interventions alter the progression of OA. More recently, platelet-rich plasma (PRP), a biological therapy, has become an emerging treatment option to improve the status of the joint for patients with OA.

PRP is an autologous blood product that is injected into the knee joint, which contains an elevated concentration of platelets above that of whole blood. However, the optimal PRP preparation is still unknown. Studies are needed that investigate optimal platelet count and how that is related to clinical outcome.

This study is designed as a double-blind randomized controlled study, where enrolled subjects are randomized to one of five treatment groups (in blocks of 10):

1. a total PRP injection dose of less than 5 billion platelets;
2. a total PRP injection dose between 5 and <10 billion platelets;
3. a total PRP injection dose between 10 and <20 billion platelets;
4. a total PRP injection dose of >20 billion platelets; and
5. a saline injection control

Each patient will be asked to complete a questionnaire at baseline, 6, 12, and 26 weeks.

After patients have completed all the study questionnaires, the Investigators will pull the results from the blood analysis, so that blood composition levels can be correlated with any pain improvements that are felt. The purpose of the study is to establish if there is a relationship between the injection dosage a patient receives and knee pain level (based on the pain scores from the self-reported questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* 40-80 years of age
* Previous diagnosis of unilateral, primary osteoarthritis of the knee
* Knee pain; duration of symptoms > 4 weeks
* K-L grade 0-4

Exclusion Criteria:

* Under 40 years of age; over 80 years of age
* Bilateral knee pain
* Duration of symptoms < 4 weeks
* NSAID or clopidogrel use in the last 7 days
* High risk of a thrombotic event if discontinuing NSAID or clopidogrel for four weeks.
* Steroid use in the last 6 weeks
* Active diagnosis of leukopenia/anemia/thrombocytopenia

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-06 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline to 26 weeks post injections
  Patient reported outcome measure: Consists of 5 subscales, one of which is "Pain". A normalized score (100 indicating no pain and 0 indicating extreme pain) is calculated for this subscale.
Western Ontario and McMaster University's Osteoarthritis Index (WOMAC) | Baseline to 26 weeks post injections
  Patient-reported outcome measure: The scores for each subscale are summed up, with a possible score range of 0-20 for Pain. Higher scores indicate worse pain.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline, 6 weeks, 12 weeks, 26 weeks post injections
  The Visual Analog Scale (VAS) is a unidimensional measure of pain intensity. The scale is most commonly anchored by "no pain " (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 10).

CONTACTS AND LOCATIONS:
Overall Officials: Leon Scott, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No